CLINICAL TRIAL: NCT00926588
Title: Stepped Care to Optimize Pain Care Effectiveness (SCOPE)
Brief Title: Stepped Care to Optimize Pain Care Effectiveness
Acronym: SCOPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 07-119
Record Dates: First submitted 2009-06-18; First posted 2009-06-23 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-07

CONDITIONS: Pain
Keywords: Pain; Telecare; Collaborative care
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stepped Care (Experimental): Patients received automated pain monitoring. A nurse care manager partnering with a physician pain specialist decide on treatment changes collaborating with primary care physicians. Structured algorithms for stepped care analgesic management and explicit decision rules for adjusting treatment are used.
  Interventions: Drug: Stepped care
- Usual Care (No Intervention): Patients receive usual care for pain from their primary care physician

INTERVENTIONS:
Drug: Stepped care — Structured algorithms for stepped care analgesic management and explicit decision rules for adjusting treatment are new tools developed for this study.
  Other Names: Optimized analgesics with collaborative care management
  Arms: Stepped Care

SUMMARY:
Pain is the most common physical symptom in primary care, accounting for an enormous burden in terms of patient suffering, quality of life, work and social disability, and health care and societal costs. Pain is particularly prevalent among veterans. Four major barriers to optimal care include underdetection of pain, inadequate initial treatment, failure to monitor adherence and symptom response, and failure to adjust treatment in patients not responding or intolerant of initial therapy. Therefore, we propose to conduct the Stepped Care to Optimize Pain care Effectiveness (SCOPE) study, a randomized clinical effectiveness trial in primary care.

DETAILED DESCRIPTION:
SCOPE will enroll 250 primary care veterans with persistent (3 months or longer) musculoskeletal pain of moderate severity, and randomize them to either the stepped care intervention or usual care control group. The intervention will be based upon the empirically-validated Three-Component Model which in SCOPE will involve collaboration between the primary care physician, a nurse pain care manager, and a supervising physician pain specialist. SCOPE will involve a telemedicine approach coupling automated home-based symptom monitoring with telephone-based nurse care management. The intervention will consist of optimized analgesic management using a stepped care approach to drug selection, symptom monitoring, dose adjustment, and switching or adding medications. All subjects will undergo comprehensive outcome assessment at baseline, 1, 3, 6 and 12 months by interviewers blinded to treatment group. Our principal aim is to test whether SCOPE is more effective than usual care in reducing pain as measured by the Brief Pain Inventory. Secondarily, we will test the impact on other pain outcomes (e.g., severity, self-efficacy, use of self-management strategies), emotional functioning, health-related quality of life, and treatment satisfaction.

ELIGIBILITY:
Inclusion Criteria:

SCOPE will enroll 250 primary care veterans with persistent (3 months or longer) musculoskeletal pain of moderate severity and randomize them to either the stepped care intervention or usual care control group.

Exclusion Criteria:

Individuals who:

* have filed a pain-related disability claim in the last 6 months;
* do not speak English;
* have moderately severe cognitive impairment;
* have schizophrenia, bipolar disorder, or other psychosis;
* are actively suicidal;
* have current illicit drug use; or
* have an anticipated life expectancy of less than 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-10; Primary Completion 2013-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Kroenke, MD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Kroenke K, Krebs E, Wu J, Bair MJ, Damush T, Chumbler N, York T, Weitlauf S, McCalley S, Evans E, Barnd J, Yu Z. Stepped Care to Optimize Pain care Effectiveness (SCOPE) trial study design and sample characteristics. Contemp Clin Trials. 2013 Mar;34(2):270-81. doi: 10.1016/j.cct.2012.11.008. Epub 2012 Dec 8. PMID 23228858
- [Result] Kroenke K, Outcalt S, Krebs E, Bair MJ, Wu J, Chumbler N, Yu Z. Association between anxiety, health-related quality of life and functional impairment in primary care patients with chronic pain. Gen Hosp Psychiatry. 2013 Jul-Aug;35(4):359-65. doi: 10.1016/j.genhosppsych.2013.03.020. Epub 2013 Apr 29. PMID 23639186
- [Result] Chumbler NR, Kroenke K, Outcalt S, Bair MJ, Krebs E, Wu J, Yu Z. Association between sense of coherence and health-related quality of life among primary care patients with chronic musculoskeletal pain. Health Qual Life Outcomes. 2013 Dec 26;11:216. doi: 10.1186/1477-7525-11-216. PMID 24369044
- [Result] Kroenke K, Krebs EE, Wu J, Yu Z, Chumbler NR, Bair MJ. Telecare collaborative management of chronic pain in primary care: a randomized clinical trial. JAMA. 2014 Jul 16;312(3):240-8. doi: 10.1001/jama.2014.7689. PMID 25027139
- [Derived] He A, Kroenke K, Stump T, Monahan PO, Connors J, Chernyak Y, Musey P. The patient health questionnaire somatization-anxiety-depression scale: Validation of the PHQ-SAD in 4 clinical trials. J Affect Disord. 2026 Apr 1;398:120906. doi: 10.1016/j.jad.2025.120906. Epub 2025 Dec 21. PMID 41436014
- [Derived] Kroenke K, Wu J, Yu Z, Bair MJ, Kean J, Stump T, Monahan PO. Patient Health Questionnaire Anxiety and Depression Scale: Initial Validation in Three Clinical Trials. Psychosom Med. 2016 Jul-Aug;78(6):716-27. doi: 10.1097/PSY.0000000000000322. PMID 27187854
- [Derived] Outcalt SD, Kroenke K, Krebs EE, Chumbler NR, Wu J, Yu Z, Bair MJ. Chronic pain and comorbid mental health conditions: independent associations of posttraumatic stress disorder and depression with pain, disability, and quality of life. J Behav Med. 2015 Jun;38(3):535-43. doi: 10.1007/s10865-015-9628-3. Epub 2015 Mar 19. PMID 25786741
- [Derived] Kroenke K, Yu Z, Wu J, Kean J, Monahan PO. Operating characteristics of PROMIS four-item depression and anxiety scales in primary care patients with chronic pain. Pain Med. 2014 Nov;15(11):1892-901. doi: 10.1111/pme.12537. Epub 2014 Aug 19. PMID 25138978

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from June 2010 through May 2012. Patients and physicians in 5 primary care clinics in the Roudebush Veterans Administration Medical Center in Indianapolis participated.
Period: Overall Study
Arm/Group | Stepped Care | Usual Care
Started | 124 | 126
Completed | 116 | 122
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stepped Care | Usual Care | Total
Number analyzed (Participants) | 124 | 126 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 124 | 126 | 250
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 28 | 43
  Male | 109 | 98 | 207
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 17 | 48
  White | 89 | 103 | 192
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 124 | 126 | 250

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory (Pain)
Description: The full scale name is the Brief Pain Inventory. This 11-item scale measures self-reported pain severity and interference. It consists of 4 pain severity items and 7 pain interference items. Each item is scored from 0 (no pain) to 10 (worse pain imaginable). There is a pain severity score (average of 4 pain severity items), pain interference score (average of 7 pain interference items), and total pain score (average of all 11 items). For all 3 scores, 0 represents the best score (i.e., least pain) and 10 represents the worst score (i.e., greatest pain).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Care | Usual Care
Number analyzed (Participants) | 124 | 126
units on a scale | 3.57 (2.22) | 4.59 (2.13)

ADVERSE EVENTS:
Arm/Group | Stepped Care | Usual Care
Serious Adverse Events (participants affected / at risk) | 22/124 | 8/126
Other Adverse Events (participants affected / at risk) | 0/124 | 0/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stepped Care (N=124) | Usual Care (N=126)
Pneumonia hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Hospitalization unrelated to research study.
Gall bladder removal surgery (Gastrointestinal disorders) | 0 | 1 — Surgery unrelated to participation in study.
Cardiac hospitalization (Cardiac disorders) | 5 | 1 — Cardiac hospitalization unrelated to participation in study.
Hospitalization due to infection (Infections and infestations) | 2 | 0 — Hospitalization not related to participation in study.
TIA hospitalization (Nervous system disorders) | 0 | 1 — Hospitalization unrelated to participation in study.
Stress center hospitalization (Psychiatric disorders) | 0 | 1 — Hospitalization unrelated to participation in study.
Sinus surgery hospitalization (Surgical and medical procedures) | 0 | 1 — Subject admitted to hospital for planned sinus surgery.
Hospitalization due to renal failure (Renal and urinary disorders) | 1 | 0 — Hospitalization unrelated to participation in study.
Hospitalization due to knee replacement (Musculoskeletal and connective tissue disorders) | 3 | 0 — Hospitalization and surgery unrelated to participation in study.
Hospitalization due to motor vehicle accident (Injury, poisoning and procedural complications) | 1 | 0 — Hospitalization unrelated to participation in study.
Bladder repair surgery and hospitalization (Renal and urinary disorders) | 1 | 0 — Surgery and hospitalization unrelated to participation in study.
Hospitalization due to removal of fibroids (Surgical and medical procedures) | 1 | 0 — Hospitalization unrelated to participation in study.
Hospitalization due to planned hysterectomy (Reproductive system and breast disorders) | 1 | 0 — Surgery and hospitalization unrelated to participation in study.
Hospitalization due to appendicitis (Gastrointestinal disorders) | 1 | 0 — Hospitalization unrelated to participation in study.
Hospitalization due to esophagogastrectomy (Gastrointestinal disorders) | 1 | 0 — Hospitalization unrelated to participation in study.
Hospitalization due to hypotension, headache, muscle ache (General disorders) | 1 | 0 — Hospitalization unrelated to participation in study.
Mental Health referral due to suicidality (Psychiatric disorders) | 0 | 1 — Unrelated to participation in study.
Hospitalization due to coronary artery bypass surgery (Cardiac disorders) | 2 | 0 — Hospitalization unrelated to participation in research study.
Subject suicidal ideation (Psychiatric disorders) | 0 | 1 — Subject revealed suicidal ideation during screening. Unrelated to participation in research study.
Death (General disorders) | 1 | 0 — Death unrelated to participation in study.
Hospitalization due to sepsis (Injury, poisoning and procedural complications) | 1 | 0 — Hospitalization unrelated to participation in research

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes